CLINICAL TRIAL: NCT05895838
Title: The Danish Out-of-Hospital Cardiac Arrest Study - a Randomized, Placebo-controlled, Double-blind, Multi Center Trial
Brief Title: The Danish Out-of-Hospital Cardiac Arrest Study
Acronym: DANOHCA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Christian Hassager (Other)
Responsible Party: Sponsor-Investigator, Christian Hassager, Professor, MD, DMSc, FESC, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-21077461; 2021-005876-21 (EudraCT Number)
Record Dates: First submitted 2023-05-10; First posted 2023-06-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome
Keywords: Out-Of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome; Systemic Inflammatory Response Syndrome; Inflammation; Cerebral perfusion; Sedation; Delirium
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome; Systemic Inflammatory Response Syndrome; Inflammation; Delirium | interventions — Dexamethasone; Olanzapine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 fashion to receive either the experimental intervention or placebo/control intervention for each of the four interventions with an assumption of no interaction.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacological interventions will be placebo controlled, and participants, care providers, investigators, and outcome assessors are blinded.
  The physiological interventions of early wakeup and extubation as well as the back-rest position are open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Dexamethasone intervention, active (Experimental): As soon as possible after hospital admittance 20 mg of dexamethasonephosphate (Dexavit, Vital Pharma Nordic ApS, Denmark) will be given intravenously (i.v.) over 15 minutes - followed by 20 mg dexamethasonephosphate (or placebo) i.v. administered daily at 0600 (or at least 8 hours after initial dose) for two days, for a total of 3 doses.
  For this arm the dexamethasonephosphate solution is provided in the "DANOHCA trial kit" in the form of Dexavit at a concentration of 4mg/mL stored in glass vials of 5mL; three vials are provided in total.
  Interventions: Drug: Dexamethasone
- Dexamethasone intervention, placebo (Placebo Comparator): As soon as possible after hospital admittance placebo (isotonic saline) will be given intravenously (i.v.) over 15 minutes - followed by placebo solution administered i.v. daily at 0600 (or at least 8 hours after initial dose) for two days, for a total of 3 doses.
  For this arm the placebo solution is provided in the "DANOHCA trial kit" in the form of isotonic sodium chloride stored in glass vials of 5mL; three vials are provided in total.
  Interventions: Drug: Dexamethasone
- Backrest elevation intervention, elevation to 35 degrees (Experimental): As soon as possible after hospital admittance the patients will have their headrest positioned at 35 degrees straight elevation of backrest in Semi-Fowler's position (elevated lower limp position). This position will be maintained during the initial 72 hours or until extubated. Adherence to assigned stratum will be checked every 8 hours and cuff pressure will be assessed and corrected if needed at the same time during the intervention period. The backrest position intervention may be temporarily canceled by the treating physician if needed for procedures or mobilization but will return to the assigned position if invasive ventilator treatment with orotracheal intubation is continued. The intervention will be terminated if the patient is extubated, or a tracheostomy is performed, during the intervention period of 72 hours.
  Interventions: Procedure: Backrest elevation
- Backrest elevation intervention, elevation to 5 degrees (Active Comparator): As soon as possible after hospital admittance the patients will have their headrest positioned at 5 degrees straight elevation of backrest in Semi-Fowler's position. This position will be maintained during the initial 72 hours or until extubated. Adherence to assigned stratum will be checked every 8 hours and cuff pressure will be assessed and corrected if needed at the same time during the intervention period. The backrest position intervention may be temporarily canceled by the treating physician if needed for procedures or mobilization but will return to the assigned position if invasive ventilator treatment with orotracheal intubation is continued. The intervention will be terminated if the patient is extubated, or a tracheostomy is performed, during the intervention period of 72 hours.
  Interventions: Procedure: Backrest elevation
- Early wake-up intervention, wake-up ≤6 hours after ICU admission (Experimental): Patients will be subjected to a wakeup call and potential extubation after ≤6 hours after admission to the ICU. Definition for "ready for extubation" will be: GCS≥12, RASS 0- -1, able to raise arm or voluntary hand shake on command, spontaneous breathing trial and low ventilator settings (pressure support≤14, PEEP≤8 (10 if obese), and FiO2≤40%). A wakeup call may be aborted for the following reasons: seizures, respiratory distress, shock, or "other cause" with specification. Sedation prior to the scheduled wakeup calls is permitted in this early wakeup call group as needed for clinical care, while it is mandatory for the late wakeup call group. For both groups sedation as needed for clinical care will be permitted after the scheduled wakeup calls.
  For this arm, information on the assigned time for wakeup call is provided in the "DANOHCA trial kit". The assigned time for wakeup will be noted in the electronic patient file.
  Interventions: Procedure: Early wakeup call
- Early wake-up intervention, wake-up 28-36 hours after ICU admission (Active Comparator): Patients will be subjected to a wakeup call and potential extubation after 28-36 hours after admission to the ICU. Definition for "ready for extubation" will be: GCS≥12, RASS 0- -1, able to raise arm or voluntary hand shake on command, spontaneous breathing trial and low ventilator settings (pressure support≤14, PEEP≤8 (10 if obese), and FiO2≤40%). A wakeup call may be aborted for the following reasons: seizures, respiratory distress, shock, or "other cause" with specification. Sedation prior to the scheduled wakeup calls is mandatory for this late wakeup call group. For both groups sedation as needed for clinical care will be permitted after the scheduled wakeup calls.
  For this arm, information on the assigned time for wakeup call is provided in the "DANOHCA trial kit". The assigned time for wakeup will be noted in the electronic patient file.
  Interventions: Procedure: Early wakeup call
- Olanzapine intervention, active (Experimental): As soon as possible after arriving at the ICU olanzapine 10mg (dissolved tablet) is administered by feeding tube. Thereafter 10 mg olanzapine is administered by feeding tube (or orally in awake patients) the following two evenings at 1800 (with a minimum of 12 hours between the initial doses) for a total of 3 doses. Due to the potential QT-prolonging effect, and concern for arrythmia, patients will be excluded prior to randomization if Long QT Syndrome (LQTS) is suspected, and telemetry of heart rhythm is mandatory for 96 hours or until life sustaining therapies are withdrawn. In case of delirium patients are treated according to standard care most often including dexmedetomidine, haloperidol or midazolam.
  For this arm the olanzapine tablets are provided in the "DANOHCA trial kit" in the form of olanzapin 10mg tablets (Accord Healthcare B.V., The Netherlands); three tablets are provided in total. Prior to administration by feeding tube the tablets are dissolved in water.
  Interventions: Drug: Olanzapine
- Olanzapine intervention, placebo (Placebo Comparator): As soon as possible after arriving at the ICU a placebo tablet (dissolved) is administered by feeding tube. Thereafter placebo will be administered by feeding tube (or orally in awake patients) the following two evenings at 1800 (with a minimum of 12 hours between the initial doses) for a total of 3 doses. Due to the potential QT-prolonging effect of olanzapine, and accompanying concern for arrythmia, patients will be excluded prior to randomization if LQTS is suspected, and telemetry of heart rhythm is mandatory for 96 hours or until life sustaining therapies are withdrawn. In case of delirium patients are treated according to standard care most often including dexmedetomidine, haloperidol or midazolam.
  For this arm the placebo tablets are provided in the "DANOHCA trial kit" in the form of placebo tablets manufactured by the Pharmacy of the Capital Region; three tablets are provided in total. Prior to administration by feeding tube the tablets are dissolved in water.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Dexamethasone — Patients will be allocated to intravenous administration of dexamethasonephosphate 20mg (Dexavit, Vital Pharma Nordic ApS, Denmark) or placebo at admission and again the following two mornings until discharge from ICU or a maximum of 3 doses.
  Other Names: Dexavit
  Arms: Dexamethasone intervention, active; Dexamethasone intervention, placebo
Procedure: Backrest elevation — Patients will be allocated to have their headrest positioned at 35 degrees backrest vs 5 degrees straight elevation of backrest for 72 hours (or until extubation if occuring prior to 72 hours).
  Arms: Backrest elevation intervention, elevation to 35 degrees; Backrest elevation intervention, elevation to 5 degrees
Procedure: Early wakeup call — Patients will be allocated to early wakeup call and potential extubation after ≤6 hours or late wakeup call and extubation between 28-36 hours after admission to the ICU.
  Arms: Early wake-up intervention, wake-up 28-36 hours after ICU admission; Early wake-up intervention, wake-up ≤6 hours after ICU admission
Drug: Olanzapine — Patients will be allocated to olanzapine 10 mg (Olanzapin, Accord Healthcare B.V., The Netherlands) administered by feeding tube (or orally in awake patients) or matching placebo at admission and again the following two evenings until discharge from ICU or a maximum of 3 doses.
  Arms: Olanzapine intervention, active; Olanzapine intervention, placebo

SUMMARY:
After resuscitation from Out-of-Hospital Cardiac Arrest (OHCA) patients experience Post Cardiac Arrest Syndrome due to ischemia and reperfusion injury. It consists of systemic inflammation, cerebral and myocardial dysfunction, and the condition that led to the arrest. Most OHCA patients will receive critical care intubated in an Intensive Care Unit (ICU). Despite this ~50% die; mainly due to brain injury. Several targets can be considered for improving outcomes. To dampen systemic inflammation and optimize cerebral perfusion seem important. Deep sedation has been required for targeted temperature management (TTM) but may also be brain protective. After end of sedation, many patients have some cerebral dysfunction that may facilitate delirium.

The aim of this trial is therefore to improve treatment of comatose OHCA patients by evaluating 4 interventions in a factorial design addressing each of these targets in a randomized clinical trial:

1. Systemic inflammation: Anti-inflammatory treatment with high dose steroids (dexamethasone) or placebo.
2. Cerebral perfusion: Backrest elevation during sedation at 5 or 35 degrees.
3. Duration of sedation: Early wakeup call and potential extubation at ≤6 hours after admission or later as current standard practice at 28-36 hours.
4. Delirium: Prophylactic treatment with anti-psychotic medication (olanzapine) or placebo.

The trial is designed as a phase III trial, randomizing 1000 patients at Danish cardiac arrest centers.

The primary endpoint is 90 days all-cause mortality for the interventions targeting systemic inflammation and cerebral perfusion, while it is days alive outside of hospital within 30 days for the interventions concerning duration of sedation and delirium.

The trial has potential to improve outcomes for comatose OHCA patients - a group with a grave prognosis with currently only limited evidence-based treatments.

DETAILED DESCRIPTION:
BACKGROUND

Initially resuscitated Out-of-Hospital Cardiac Arrest (OHCA) patients admitted to a hospital are often in an unstable condition necessitating both circulatory and respiratory support. Most of these patients experiences the Post Cardiac Arrest Syndrome (PCAS) immediately after resuscitation due to a whole-body ischemia and reperfusion injury. It consists of four elements: 1) a universal systemic inflammatory response, 2) cerebral dysfunction, 3) myocardial dysfunction, and 4) the precipitation condition that led to the cardiac arrest - often a coronary occlusion.

The majority of OHCA patients have a presumed cardiac cause for their cardiac arrest. These patients are all evaluated for immediate coronary revascularization, stabilized with vasopressors, inotropes or mechanical circulatory support, and if comatose further sedated, connected to a ventilator and given targeted temperature management (TTM) for at least 24 hours. Half of the admitted resuscitated OHCA patients still die during the hospitalization despite all these interventions. The main cause of death is withdrawal of life sustaining therapy due to irreversible brain injury.

Several targets can be approached in order to potentially improve the outcome of OHCA patients. During the initial phase early after hospital admittance, interventions to dampen the systemic inflammatory response and efforts to secure optimum cerebral perfusion pressure seem intuitive important. Deep sedation has been required for TTM but may also have brain protective effects. After discontinuation of the sedation when the TTM is over, most patients have some degree of cerebral dysfunction. This may make them more prone to develop delirium in the days after awakening which is an independent risk factor in critical ill patients.

The DANOHCA trial will therefore evaluate new potential interventions to each of these different targets: systemic inflammation, cerebral perfusion, duration of sedation, and delirium.

INTERVENTIONS

High-dose steroids to dampen systemic inflammation in resuscitated OHCA patients:

By randomization, the patients will be allocated 1:1 to either dexamethasone (administered as dexamethasonephosphate) or placebo for three days. As soon as possible after admittance 20 mg of dexamethasonephosphate (Dexavit, Vital Pharma Nordic ApS, Denmark) or placebo will be given intravenously (i.v.) over 15 minutes - followed by 20 mg dexamethasonephosphate (or placebo) i.v. administered daily at 0600 (or at least 8 hours after initial dose) for two days, for a total of 3 doses.

Backrest elevation in post cardiac arrest care and outcome for OHCA patients:

By randomization, the patients will be allocated to have their headrest positioned at 5 degrees backrest vs 35 degrees straight elevation of backrest in Semi-Fowler's position (elevated lower limp position) during the initial 72 hours or until extubated. The adherence to the assigned stratum will be checked every 8 hours and cuff pressure will be assessed and corrected if needed at the same time during the intervention period. The backrest position intervention may be temporarily canceled by the treating physician if needed for procedures or mobilization but will return to the assigned position if invasive ventilator treatment with orotracheal intubation is continued. The intervention will be terminated if the patient is extubated, or a tracheostomy is performed, during the intervention period of 72 hours.

Early wake up and extubation in OHCA patients:

By randomization, the patients will be allocated 1:1 to early wakeup call and potential extubation after ≤6 hours or late wakeup call and extubation between 28-36 hours after admission to the ICU. Definition for "ready for extubation" will be: GCS≥12, RASS 0 to -1, able to raise arm or voluntary hand shake on command, spontaneous breathing trial and low ventilator settings (pressure support≤14, PEEP≤8 (10 if obese), and FiO2≤40%). A wakeup call may for both groups be aborted for the following reasons: seizures, respiratory distress, shock, or "other cause" with specification. Sedation prior to the scheduled wakeup calls is permitted in the early wakeup call group as needed for clinical care, while it is mandatory for the late wakeup call group. For both groups, sedation as needed for clinical care will be permitted after the scheduled wakeup call.

Prophylactic use of olanzapine to prevent delirium in patients resuscitated from OHCA:

By randomization, the patients will be allocated 1:1 to olanzapine 10 mg (Olanzapin, Accord Healthcare B.V., The Netherlands) administered by feeding tube (or orally in awake patients) or matching placebo at admission and again the following two evenings until discharge from ICU or a maximum of 3 doses. As soon as possible after arriving at the ICU: olanzapine/placebo is given by feeding tube. Thereafter 10 mg olanzapine or matching placebo will be given by feeding tube (or orally in awake patients) the following two evenings at 1800 (with a minimum of 12 hours between the initial doses) for a total of 3 doses. Due to the potential QT-prolonging effect, and accompanying concern for arrythmia, patients will be excluded prior to randomization if Long QT Syndrome (LQTS) has been confirmed or suspected, and all patients will be monitored by mandatory telemetry of heart rhythm for 96 hours or until life sustaining therapies are withdrawn. In case of delirium, patients are treated according to standard care most often including dexmedetomidine, haloperidol or midazolam.

STUDY DESIGN

The study is an investigator-initiated, randomized, controlled, multicenter clinical trial with co-enrollment into 4 different interventions. The pharmacological interventions are placebo-controlled, double-blind interventions and physiological interventions of early wakeup and extubation, as well as the back-rest position interventions are open label. Following successful completion of screening procedures, patients will be randomized in a 1:1 fashion to receive either the active intervention or placebo/control intervention for each intervention. The randomization will be revealed by opening a sealed box (referred to as the "DANOHCA trial kit" below) containing the study drug vials/tablets, instructions for wakeup and extubation and backrest positioning.

The trial aims to include 1000 patients from 5 sites. Approximately 350 patients are eligible for inclusion at the five hospitals combined each year, and therefore inclusion is expected to be concluded after 3-4 years.

Sub-studies further investigating the effect of the interventions will be performed. A research biobank will be established. Further co-enrollment into additional trials must be permitted by the steering group after careful assessment of risk of interaction with the four per-protocol interventions.

STATISTICAL ANALYSES

The data will be analyzed and reported as 4 individual trials, hence no adjustment for multiple comparison is planned.

Should more than one of the interventions be non-neutral a post hoc evaluation of interaction will be performed and highlighted in the reporting of the results. Also, as an investigation of potential safety aspects related to possible interactions between the four interventions, interactions related to mortality and occurrence of other SAE' will be reported.

All analyses will be conducted in the modified intention-to-treat (ITT) population with a set two-level significance level of 0.05. Modified ITT in this regard means that patients included without fulfilling the inclusion criteria will be excluded from the analyses.

Throughout, categorical variables will be presented as numbers (frequencies), whereas continuous variables will be presented as mean ±SD if normally distributed, and as median (25th percentile-75th percentile) if non-normally distributed. The primary analysis of primary endpoint will include the modified ITT population. Further the investigators plan a sensitivity analysis in the per protocol population to assess the effect. The per protocol cohort will be defined as only those trial participants who have received ALL scheduled doses of the pharmacologic interventions, have adhered to the assigned back-rest position for ≥80% of the time, and have had a wake-up call attempted within the assigned time frames.

Continuous endpoints being assessed at multiple time points will be analyzed by application of linear mixed models of covariance. The main result of these analyses will be the treatment-by-time interaction as a marker of whether the individual endpoint changes differently over time in the active intervention vs. the placebo arm, and group differences will be reported as relative differences in %. Logarithmic transformation will be applied to approximate normal distribution as appropriate.

Categorical endpoints by treatment allocation will be analyzed by the Chi-Squared or the Fisher's exact test, as appropriate.

For analysis of survival data, Kaplan-Meier curves for each allocation group will be estimated, graphically displayed, and compared by the log-rank test. Further Cox proportional hazard models will be applied to assess differences in time to death between treatment groups. These models will sequentially be adjusted for the interaction between treatment allocation, and each of the following variables: sex, age, time to ROSC, lactate level upon admission, shockable primary rhythm, witnessed cardiac arrest, bystander performed cardiopulmonary resuscitation, presence of STEMI in the admission ECG. Further, models stratified by cause of death (cardiovascular, neurological, multi-organ failure) will be applied as hypothesis generating. Any changes from the pre-specified analysis plan will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. OHCA of presumed cardiac cause
3. Sustained ROSC, defined as persistent signs of circulation and no need for chest compressions or mechanical circulatory support for 20 minutes
4. Unconsciousness (GCS <9) (patients not able to obey verbal commands) after sustained ROSC at the time of randomization

Exclusion Criteria:

1. Females of childbearing potential if pregnancy is suspected (unless a negative HCG test can rule out pregnancy within the inclusion window)
2. Known bleeding diathesis (medically induced coagulopathy (e.g. warfarin, NOAC, clopidogrel) does not exclude the patient)
3. Suspected or confirmed acute intracranial bleeding
4. Suspected or confirmed acute stroke
5. Unwitnessed asystole
6. Known limitations in therapy and Do Not Resuscitate-order
7. Known disease making 180 days survival unlikely
8. Known pre-arrest CPC 3 or 4 functional status
9. >3 hours (180 minutes) from ROSC to screening
10. Systolic blood pressure <80 mm Hg despite fluid loading/vasopressor and/or inotropic medication (If the systolic blood pressure is recovering during the inclusion window of 180 minutes the patient may be included)
11. Use of intra-aortic balloon pump/axial flow device/ECMO (If the patient is weaned and the device is removed during the inclusion window of 180 minutes the patient may be included)
12. Temperature on admission <30°C
13. Known allergy for dexamethasone or olanzapine
14. Ongoing (within 48 h) treatment with olanzapine or dexamethasone
15. Known back or hip condition that precluded the patients from being positioned with backrest from 0 to 45-degree angle
16. Known or suspected Long QT Syndrome (LQTS)
17. Known active fungal disease. Localized skin lesions do not exclude patients from inclusion
18. Estimated body weight <45kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Steroid intervention primary endpoint: All-cause mortality | 90 days
  Number of patients dying from all causes
Back rest position intervention primary endpoint: All-cause mortality | 90 days
  Number of patients dying from all causes
Early wakeup and extubation intervention primary endpoint: Days alive outside hospital | 30 days
  Counted as days alive outside of hospital after discharge
Olanzapine intervention primary endpoint: Days alive outside hospital | 30 days
  Counted as days alive outside of hospital after discharge

SECONDARY OUTCOMES:
Number of patients dying from all causes | 90 days
  Applies to the Early wakeup and extubation intervention, as well as Olanzapine intervention
Neuron Specific Enolase and Neurofilament Light Chain levels | 48 hours
  Serum markers for brain injury; Differences in levels between intervention groups assessed at 48 hours; Applies to all interventions
Troponin I, Troponin T, and Creatine Kinase Myocardial Band | 0-72 hours
  Plasma markers of myocardial injury; Differences in levels between intervention groups assessed during initial 72 hours; Applies to all interventions
Plasma Creatinine and use of dialysis | Creatinine: initial 72 hours; Dialysis: initial 30 days
  Markers of kidney injury; Creatinine will be assessed during initial 72 hours, and use of dialysis will be assessed during initial 30 days
Vasopressors and inotropic drugs | Initial ICU stay, during the first 36 hours
  Use of vasopressors and inotropic drugs in the Intensive Care Unit (ICU), characterised as cumulative doses and total doses
Mixed blood venous saturation | Assessed at 12, 24 and 36 hours and after this, once daily during initial ICU stay, up to 90 days
  Oxygen saturation assessed by blood gas analyses of blood drawn from a pulmonary artery catheter
Duration of intubation | Up to 90 days
  Assessed as the duration of intubation from randomization till extubation during initial ICU stay (oral and tracheostomy combined)
Unconsciousness | 96 hours
  Assessed as the number of unconscious patients at 96 hours
CAM-ICU positive status | 24 hours after extubation
  Assessed as the number of CAM-ICU positive patients 24 hours after extubation
CAM-ICU negative days | Up to 90 days
  Assessed as the number of CAM-ICU negative days during initial ICU stay
Pharmacological treatment for delirium | From randomization till discharge from initial ICU stay, up to 90 days
  Assessed as the number of days without pharmacological treatment for delirium (other than study drug during the intervention period)
Length of hospital stay | From randomization till discharge from hospital or in-patient rehabilitation, up to 90 days
  Assessed as the hospital length of stay (including in-patient rehabilitation and transfer to referral hospital)
Cerebral Performance Category (CPC) | Up to 6 months
  CPC score at at ICU discharge, at hospital discharge, and at ambulatory follow-up (scheduled visit at 3 to 6 months after the cardiac arrest). The CPC score ranges from 1 to 5 with higher scores indicating worse outcomes.
modified Rankin Scale (mRS) | Up to 6 months
  mRS score at at ICU discharge, at hospital discharge, and at ambulatory follow-up (scheduled visit at 3 to 6 months after the cardiac arrest). The mRS score ranges from 0 to 6 with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hassager, MD DMSc, Study Chair — Dept. of Cardiology, Rigshospitalet; Jesper Kjaergaard, MD PhD DMSc, Principal Investigator — Dept. of Cardiology, Rigshospitalet
Locations (5):
- Denmark (5):
  - Dept. of Cardiology, The Heart Centre, Copenhagen University Hospital Rigshospitalet, Copenhagen, Capital Region of Denmark
  - The Department of Intensive Care, Aalborg University Hospital, Aalborg
  - The Department of Intensive Care, Aarhus University Hospital, Aarhus
  - Department of Anaesthesiology and Intensive Care Medicine, Zealand University Hospital, Køge
  - The Department of Cardiothoracic Anaesthesiology, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No